CLINICAL TRIAL: NCT05654402
Title: Non-invasive Measurement of Arterial Stiffness by Pulse Wave Velocity.
Brief Title: Non-invasive Measurement of Arterial Stiffness
Acronym: NIVOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); M3DISIM (Other)
Responsible Party: Sponsor
Other Study IDs: APHP2203812
Record Dates: First submitted 2022-11-21; First posted 2022-12-16 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia, Local; Anesthesia
Keywords: Predictive medicine; Pulse wave velocity; Cardiovascular complications; Predictive Biomarker; Arterial stiffness
MeSH Terms: interventions — Pulse Wave Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Non-invasive measurement of carotid-femoral transit time by Doppler velocimetry (Athys Medical©) - WAKIe R3 2TC®) (PWV in cm/s) — * Measurement of the carotid-femoral transit time (ms) (recorded on Data Warehouse Connect).
  * Measurement of the distance between the carotid and femoral points with a tape measure (m).
  * Calculation of the propagation speed of the wave PWV (expressed in m/s).
  For all patients PWV in (m/s=) will be collected over three distinct periods:
  * Before induction (awake without premedication)
  * During general anesthesia or loco-regional anesthesia
  * Upon awakening from general anesthesia or lifting of the loco-regional anaesthesia

SUMMARY:
Reducing the risk of perioperative cardiovascular complications is a major issue for anesthesiology practice and research. Carotid-Femoral Pulse Wave Velocity (PWVcf)is a predictive, early and independent biomarker of cardiovascular events. Despite the unanimous support for PWVcf, it has not been widely used in routine clinical practice because of the complexity of the measurement method. Our team has developed a method to estimate PWVcf continuously in the operating room from the data obtained by the usual monitoring: an electrocardiogram (ECG), a digital photoplethysmography (PPG) and an oscillometric brachial sphygmomanometer for non-invasive blood pressure measurement (NIP). The objective of this study is to validate, during anesthesia, the method of estimation of PWV (obtained using the usual monitoring tools including the parameters derived from the SpO2 signal, NIBP and ECG) by comparing it to the reference method by measuring the carotid-femoral transit time obtained by Doppler effect. The measurement of the carotid-femoral transit time obtained by Doppler effect is totally non-invasive.

DETAILED DESCRIPTION:
Reducing the risk of perioperative cardiovascular complications is a major issue for anesthesiology practice and research. The risk of postoperative cardiovascular complications could therefore be stratified by screening "rigid" patients who have no cardiovascular risk factors.

Assessment of large-caliber artery stiffness is a predictive, early, and independent biomarker of cardiovascular events, currently included in European guidelines for the management of hypertension. It is also a physiological parameter that reflects left ventricular afterload and is very useful during the management of patients under general anesthesia. The parameter considered as the "gold standard" for the evaluation of this arterial stiffness is the measurement of the pulse wave velocity (PWV) or carotid-femoral pulse wave velocity (PWVcf). PWVcf is the propagation speed of the pulse wave from the carotid artery to the femoral artery, i.e., the time it takes for the pulse wave to travel from a point in the carotid artery to a point in the femoral artery. PWVcf has not become widespread in routine clinical practice because of the complexity of the measurement method. Indeed, PWVcf measurement can only be performed by imaging (MRI), or by ultrasound technique (combined carotid and femoral Doppler) or by combined tonometry (e.g. SphygmoCor, Complior). These techniques require specific equipment as well as training, expertise and learning of the collection technique. Previous studies have allowed the development of an algorithm allowing indirect measurement of PWV from combined carotid-femoral Doppler and tonometry PWVcf measurements in patients under general anesthesia. Thanks to the acquisition tools, the data will be available and of high quality, guaranteeing that the tools/algorithm developed from them will not be biased and will be more efficient.

The objective of this study is to validate, during anesthesia, the method of estimation of PWV (obtained using the usual monitoring tools including the parameters derived from the SpO2 signal, NIBP and ECG) by comparing it to the reference method by measuring the carotid-femoral transit time obtained by Doppler effect.

Patients over 18 years old are eligible to participate in this protocol. During the anaesthesia consultation, patients will be given a letter of information on the objectives and progress of the study. Their non-objection to participate in this study will be collected at the latest during the pre-anesthetic visit, the day before the operation, after a period of reflection.

The protocol will start on the day of the operation. The procedures will be performed under general anesthesia or locoregional anesthesia. The protocol does not interact with the care procedure.

The 2 self-adhesive Doppler sensors are placed at the level of the common carotid and superficial femoral arteries at the level of the Scarpa. The visualized signal is automatically validated after several cycles when the quality is satisfactory (Athys Medical©) - WAKIe R3 2TC®). This signal, allowing the measurement of the carotid-femoral transit time, is then recorded on Data Warehouse Connect.

The distance between the two measurement points is measured with a tape measure. Knowing the carotid-femoral transit time, the propagation speed of the wave (expressed in m/s) can be calculated.

No invasive devices are used in addition to those required for anesthesia. All the monitoring instruments described above, except the one studied, are already used routinely in our department. The duration of anesthesia is not prolonged for the study. The Doppler is performed during the awake, anesthetic induction and awake phase.

No additional exams will be performed. The anesthetic strategy is decided by the anesthesiologist in charge of the operation.

The physician in charge of the study collecting the data does not participate at any time in the management of the patient. The measures cannot influence the prescribing physician since at this stage the data are not yet analyzed and available

The estimation of the number of subjects to be included is based on the primary endpoint, namely the intraclass correlation coefficient. Thus, to demonstrate an ICC of 0.9 with a confidence interval of 0.1, for a 5% alpha risk, it is necessary to include 98 patients.

Continuous data are expressed as median [interquartile] and categorical data as n (%). Categorical variables will be compared by Mann-Whtney test and continuous variables by Wilcoxon test.

The agreement between the two methods will be evaluated by the intra-class correlation coefficient as well as by the Bland-Altman representation (with determination of the bias and the limits of agreement), for the different parameters of interest. All statistical analyses will be performed using R statistical software (The 'R' Foundation for Statistical Computing, Vienna, Austria). The results will be expressed as means (± standard deviation). A p-value less than 0.05 is considered significant

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age ( 18 years)
* Eligible for a scheduled surgical procedure under general or locoregional anesthesia.
* Patients who have expressed no objection to participating in this research

Exclusion Criteria:

* Patients under 18 years of age.
* Carotid or femoral space not available
* Atrial fibrillation arrhythmia (AFA)
* Advanced obliterative arteriopathy of the lower limbs (grade III and IV - Leriche and Fontaine)
* Patient opposed to participation in the protocol
* Pregnant woman
* Patient under judicial protection
* Patient not affiliated to a social health system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants or populations are selected based on predefined criteria.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
To study the concordance of carotid-femoral pulse wave velocity (PWVcf) values obtained by carotid-femoral Doppler method with those obtained completely noninvasively by continuous PWV estimation under the same conditions during anesthesia. | 1 day
  Non-invasive measurement of carotid-femoral transit time by Doppler velocimetry (PWV in cm/s).
Study concordance of carotid-femoral pulse wave velocity values obtained by carotid-femoral Doppler method and those obtained completely noninvasively by continuous PWV estimation under the same conditions during anesthesia using mean arterial pressure | 1 day
  Non-invasive continuous measurement of mean arterial pressure in mmHg.
To study the concordance of carotid-femoral pulse wave velocity values obtained by carotid-femoral Doppler method with those obtained completely noninvasively by continuous PWV estimation under the same conditions during anesthesia using blood pressure. | 1 day
  Discontinuous measurement of blood pressure with an oscillometric brachial blood pressure monitor.
To study the concordance of carotid-femoral pulse wave velocity (PWVcf) values obtained by carotid-femoral Doppler method with those obtained completely noninvasively by continuous PWV estimation under the same conditions during anesthesia using ECG. | 1 day
  Continuous ECG recording.
Study concordance of carotid-femoral pulse wave velocity values obtained by carotid-femoral Doppler method and those obtained by continuous PWV estimation under the same conditions during anesthesia thanks to digital photoplethysmography recording | 1 day
  Continuous digital photoplethysmography recording exprimed in %.
Study concordance of carotid-femoral pulse wave velocity values obtained by carotid-femoral Doppler method and those obtained completely noninvasively by continuous PWV estimation under the same conditions during anesthesia thanks to administred agents | 1 day
  Quantification of delivered doses of hypnotics, morphinics and paralytic agents.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim MD MATEO, Study Director — Assistance Publique - Hôpitaux de Paris; Fabrice MD VALLEE, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris, Department of Anesthesiology and Intensive Care
Locations (1):
- AP-HP, Lariboisière Hospital, Department of Anesthesiology and Intensive Care, Paris, France